CLINICAL TRIAL: NCT03610360
Title: A Randomized, Open-Label Phase II/III Study With Dendritic Cells Loaded With Allogeneic Tumour Cell Lysate (PheraLys) in Subjects With Mesothelioma as Maintenance Treatment (MesoPher) After Chemotherapy
Brief Title: DENdritic Cell Immunotherapy for Mesothelioma
Acronym: DENIM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amphera BV (Industry)
Collaborators: TMC Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM04; DENIM (Other: Amphera)
Record Dates: First submitted 2018-07-24; First posted 2018-08-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Mesothelioma
Keywords: DENIM
MeSH Terms: conditions — Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Arm A will receive the study drug MesoPher plus best supportive care
  Interventions: Drug: MesoPher
- Arm B (No Intervention): Arm B will follow best supportive care as deemed appropriate by the investigator.

INTERVENTIONS:
Drug: MesoPher — Subjects in Arm A will undergo leukapheresis to obtain monocytes from which dendritic cells will be generated. These dendritic cells will be loaded in vitro with an allogeneic tumor cell lysate (PheraLys). Treatment with autologous dendritic cells loaded with PheraLys is called MesoPher
  Arms: Arm A

SUMMARY:
This study is to evaluate the overall survival (OS) rate (determined from the time of randomization in the study) of subjects who receive dendritic cell immunotherapy with MesoPher plus best supportive care (BSC) compared to BSC alone.

DETAILED DESCRIPTION:
This is an open-label, randomized Phase II/III study in adult subjects with mesothelioma to evaluate the efficacy and anti-tumor activity of dendritic cell immunotherapy with MesoPher plus best supportive care compared to best supportive care alone. The safety, tolerability, quality of life and immunogenicity of MesoPher will also be evaluated.

The study includes a screening phase, a 7 month open-label treatment phase during which subjects visit the study center for administration of study drug and follow-up evaluations. An end-of-study (EoS) visit will be performed after completion of the study, after which data on survival, subsequent therapies and response to these therapies will be collected.

A target of 230 subjects satisfying all study criteria, will be randomized to receive either dendritic cell therapy plus best supportive care (Arm A) or best supportive care alone (Arm B).

Subjects in Arm A will undergo leukapheresis to obtain monocytes from which dendritic cells will be generated. These dendritic cells will be loaded in vitro with an allogeneic tumor cell lysate (PheraLys). Treatment with autologous dendritic cells loaded with PheraLys is called MesoPher. The treatment with Mesopher will start within 9 to 13 weeks after the last dose of chemotherapy. Subjects will receive 3 bi-weekly injections with MesoPher in addition to BSC. In case of stable disease or partial/complete response, an additional 2 injections will be given at weeks 18 and 30. Subjects will be administered with a maximum of 5 doses of MesoPher.

Subjects in Arm B will be treated with best supportive care according to the discretion of the local investigator.

ELIGIBILITY:
Subjects will only be included with a histologically confirmed diagnosis of pleural malignant mesothelioma, who are non-progressive after 4 to 6 cycles with first line chemotherapy with antifolate/platinum.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | from randomisation to study end (the last visit for the last subject participating in the study and the last data collection point completed) assessed in up to 102 weeks
  The primary outcome measure of this study is to evaluate the overall survival (OS) rate of subjects who receive dendritic cell immunotherapy with MesoPher plus best supportive care (BSC) compared to BSC alone. Overall survival rate will be determined from randomisation until death.

CONTACTS AND LOCATIONS:
Locations (6):
- University Hospital Antwerp, Antwerp, Belgium
- Centre Hospitalier Régional Universitaire de Lille, Lille, France
- Universitá Politecnica delle Marche - Ospedali Riuniti di Ancona, Ancona, Italy
- Netherlands (2):
  - Netherlands Cancer Institue, Amsterdam
  - Erasmus Medical Centre, Rotterdam
- University of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aerts JG, Belderbos R, Baas P, Scherpereel A, Bezemer K, Enninga I, Meijer R, Willemsen M, Berardi R, Fennell D, Kerstens R, Cornelissen R, van Meerbeeck JP; DENIM team. Dendritic cells loaded with allogeneic tumour cell lysate plus best supportive care versus best supportive care alone in patients with pleural mesothelioma as maintenance therapy after chemotherapy (DENIM): a multicentre, open-label, randomised, phase 2/3 study. Lancet Oncol. 2024 Jul;25(7):865-878. doi: 10.1016/S1470-2045(24)00191-8. Epub 2024 Jun 4. PMID 38848742